CLINICAL TRIAL: NCT02569866
Title: Antibiotics After Breast Reduction:Clinical Trial With Randomization
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Collaborators: Universidade do Vale do Sapucai (Other)
Responsible Party: Principal Investigator, Edgard da Silva Garcia, Edgard da Silva Garcia, Professor, Universidade do Vale do Sapucaí, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ESG180402
Record Dates: First submitted 2015-10-04; First posted 2015-10-07 (Estimated); Last update posted 2018-04-20 (Actual); Status verified 2018-04

CONDITIONS: Surgical Site Infection
Keywords: plastic surgery; mammaplasty; wound infection; prophylaxis
MeSH Terms: conditions — Surgical Wound Infection; Wound Infection | interventions — Cephalexin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Antibiotics Group (Active Comparator): Capsules containing cephalexin/500mg will be administrated to the subjects, 4 times daily, for seven days during the postoperative period of reduction mammaplasty.
  Interventions: Drug: Cephalexin
- Placebo Group (Placebo Comparator): Capsules containing placebo/500mg will be administrated to the subjects, 4 times daily, for seven days during the postoperative period of reduction mammaplasty.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cephalexin — Capsules containing cephalexin/500mg
  Arms: Antibiotics Group
Drug: Placebo — Capsules containing placebo/500mg
  Arms: Placebo Group

SUMMARY:
This study was designed to determine the role of antibiotics reduction mammaplasty influence surgical site infections rates.

DETAILED DESCRIPTION:
Prevention of SSI is important due to its morbidity, longer hospital stays and higher costs. In many surgical procedures where the risk of infection is relatively low and the postoperative infection can be treated properly, the role of antibiotics is not clear.

Despite the lack of evidence from prospective randomized controlled trials of evaluation, the use of antibiotics in plastic surgery is widespread in order to offer the highest safety standards patients.

The breast reduction is defined as "clean surgery" with a lower infection rate to 3.4%. Thus, the antibiotic is not recommended. However, studies have shown a real rate of infection associated with procedures ranging from 4-36%.

Thus, this trial was designed to verify the role of antibiotics in reduction mammaplasty.

ELIGIBILITY:
Inclusion Criteria:

* Breast hypertrophy
* Body mass index between 19 to 30 kg/m2

Exclusion Criteria:

* Patients undergoing a surgical procedure in the breast
* Diagnosis of breast pathology
* Smoking
* Childbirth or lactation less than a year
* Uncontrolled comorbidities
* Use of immunosuppressive drugs
* Misuse of capsules supplied
* Absence during the weekly follow-up

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 124 (Actual)
Dates: Start 2014-11; Primary Completion 2016-05 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Surgical site infection in the postoperative of reduction mammaplasty. | 30 days postoperatively
  After surgery, the patients will be followed for 30 days and surgical site infection rates will be observed in both groups, according to the CDC criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Lydia M Ferreira, PhD, Study Chair — Federal University of São Paulo
Locations (1):
- Hospital das Clínicas Samuel Libanio, Pouso Alegre, Minas Gerais, Brazil

REFERENCES:
- [Background] Veiga-Filho J, Veiga DF, Sabino-Neto M, Amorim MC, Novo NF, Ferreira LM. The role of antibiotics in reduction mammaplasty. Ann Plast Surg. 2010 Aug;65(2):144-6. doi: 10.1097/SAP.0b013e3181c47d88. PMID 20585232
- [Derived] Garcia ES, Veiga DF, Veiga-Filho J, Cabral IV, Pinto NL, Novo NF, Sabino Neto M, Ferreira LM. Antibiotic prophylaxis in reduction mammaplasty: study protocol for a randomized controlled trial. Trials. 2016 Nov 30;17(1):567. doi: 10.1186/s13063-016-1700-y. PMID 27899130